CLINICAL TRIAL: NCT01369108
Title: Clinical Evaluation of a Low Shrinkage Flowable Resin Composite in Adult Teeth
Brief Title: Clinical Study on a New Flowable Composite as a Restorative in Adult Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-10-013
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries
Keywords: small Class I; molar and premolar; low stress flowable composite; adult; Restoration; small caries lesions
MeSH Terms: conditions — Dental Caries; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flowable composite (Experimental): Flowable composite
  Interventions: Device: Flowable composite
- Conventional composite (Active Comparator): Highly filled conventional composite restorative
  Interventions: Device: Conventional composite restorative

INTERVENTIONS:
Device: Flowable composite — Restoration of small Class V and I cavities in molar and premolar teeth
  Other Names: Filtek Supreme Ultra Flowable Restorative 3M ESPE)
  Arms: Flowable composite
Device: Conventional composite restorative — Restoration of small Class V and I cavities in molar and premolar teeth
  Arms: Conventional composite

SUMMARY:
Study hypothesis: a new, low polymerization stress flowable composite performs no differently to a conventional, highly filled composite filling material when used as a restorative in small cavities in back teeth.

Study will evaluate the clinical performance of a low shrinking flowable composite filling material, compared with a conventional, highly filled composite restorative when used to permanently fill small cavities in molar and premolar teeth in adult patients.

DETAILED DESCRIPTION:
The study will evaluate clinical performance of a low shrink flowable composite filling material and compare it with a conventional, highly filled composite. The study materials will be used to restore small cavities in molar and premolar teeth in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* must give written consent
* be in good general health
* be available for required follow-up visits
* have at least 28 teeth

Exclusion Criteria:

* has rampant, uncontrolled caries
* has advanced, untreated periodontal disease
* heavy use of smoking tobacco (2 packs or equivalent a day)or chewing tobacco
* has systemic or local disorders that contra-indicate the dental procedures needed in this study
* has evidence of xerostomia
* has evidence of severe bruxing or clenching, or in need of Temporomandibular Joint (TMJ) related therapy
* is pregnant at time of screening or tooth restoration
* has known sensitivity to acrylates or related materials

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John O Burgess, DDS, MS, Principal Investigator — Unversity of Alabama at Birmingam Dental School
Locations (1):
- University of Alabama at Birmingham School of Dentistry, 605 School of Dentistry Building, 1919 7th Avenue South, Birmingham, Alabama, United States

REFERENCES:
- [Result] Lawson NC, Radhakrishnan R, Givan DA, Ramp LC, Burgess JO. Two-year Randomized, Controlled Clinical Trial of a Flowable and Conventional Composite in Class I Restorations. Oper Dent. 2015 Nov-Dec;40(6):594-602. doi: 10.2341/15-038-C. Epub 2015 Aug 3. PMID 26237643

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Each enrolled patient possessed two teeth that met the inclusion criteria. Of these, 120 teeth, 60 were allocated to the comparator group (Filtek Supreme Ultra Universal restorative) and 60 were allocated to the experimental group (Filtek Supreme Ultra Flowable.
  Flowable composite: Restoration of small Class V and I cavities in molar and premolar teeth
  Conventional composite restorative: Restoration of small Class V and I cavities in molar and premolar teeth
Period: Overall Study
Arm/Group | All Participants
Started | 60 (120 teeth)
Completed | 49
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 52 [19 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Clinical Performance by Cvar & Ryge Scores
Description: Clinical performance reported on 6 parameters as the % of teeth with perfect scores ("A" rating).
  Cvar & Ryge scores measure 6 parameters: Anatomic form (rated A,B= satisfactory, C=unsatisfactory); Color Match (A=match, B=mismatch, but within normal, C=mismatch outside normal); Marginal Adaptation (A=no visible crevice, B=no exposure of dentin, C=defect to enamel-dentine junction, D= fracture, missing); Marginal Discoloration (A=none, B= marginal discoloration, C=marginal discoloration to pulpal direction); Surface Integrity (A=smooth, B=slight rough, C=Pitted, D=fracture)'Secondary caries (A=none, D=present).
Time Frame: baseline, 6, 12 and 24 months
Measure: Number; unit: percent of teeth
Units Other Than Participants: teeth
Arm/Group | Flowable Composite | Conventional Composite
Number analyzed (Participants) | 49 | 49
Number analyzed (teeth) | 49 | 49
percent of teeth
  Color match baseline | 96.6 | 88.3
  Anatomic baseline | 100.0 | 100.0
  Marginal adaptation baseline | 96.6 | 98.3
  Marginal discoloration Baseline | 98.3 | 98.3
  Surface Integrity Baseline | 98.3 | 96.7
  Secondar carries Baseline | 100. | 98.3
  Anatomic form 6 Mo | 100. | 98.3
  Color match form 6 Mo | 96.6 | 91.7
  Marginal adaptation 6 Mo | 93.2 | 88.3
  Marginal discoloration 6 Mo | 96.6 | 95.0
  Surface integrity 6 Mo | 96.6 | 90.0
  Secondary caries 6 Mo | 100. | 96.7
  Anatomic form 12 Mo | 96.4 | 94.6
  Color match 12 Mo | 92.7 | 83.9
  Marginal adaption 12 Mo | 81.8 | 78.6
  Marginal discoloration 12 Mo | 90.9 | 90.1
  Surface Integrity 12 Mo | 92.7 | 78.6
  Secondary caries 12 Mo | 94.5 | 94.6
  Anatomic form 24 Mo | 89.8 | 86.0
  Color match 24 Mo | 85.7 | 78.0
  Marginal adaption 24 Mo | 83.7 | 80.0
  Marginal discoloraton 24 Mo | 85.7 | 80.0
  Surface integrity 24 Mo | 79.6 | 78.0
  Secondary caries 24 Mo | 93.9 | 94
Statistical Analysis 1: Comparison: Flowable Composite vs Conventional Composite; null hypothesis no difference in anatomic form; Test type: Superiority or Other; p = 0.8, ANOVA
Statistical Analysis 2: Comparison: Flowable Composite vs Conventional Composite; null hypothesis no difference in margin adaptation; Test type: Superiority or Other; p = 0.89, ANOVA
Statistical Analysis 3: Comparison: Flowable Composite vs Conventional Composite; null hypothesis no difference in margin discoloration; Test type: Superiority or Other; p = 0.79, ANOVA
Statistical Analysis 4: Comparison: Flowable Composite vs Conventional Composite; null hypothesis no difference in surface integrity; Test type: Superiority or Other; p = 0.18, ANOVA
Statistical Analysis 5: Comparison: Flowable Composite vs Conventional Composite; null hypothesis no difference in secondary caries; Test type: Superiority or Other; p = 0.66, ANOVA

2. Primary Outcome: Clinical Performance by VAS (Pain Scale)
Description: Sensitivity to cold was measured by applying a cotton pellet soaked with pulp vitality refrigerant spray (Endo Ice, Coltene/ Whaledent, Cuyahoga Falls, OH, USA) to the tooth for three seconds. Sensitivity to biting was measured by having the patient bite on a cotton roll for five seconds. After each test, the subject was asked to place an ''X'' on a 10-mm line labeled ''1'' on the left and ''10'' on the right. Patients were told that a ''10'' represents the worst pain they can imagine (ie, childbirth, major surgery, or kidney stone) and that ''1'' represents no sensation at all.
Time Frame: baseline, 6, 12 and 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: teeth
Arm/Group | Flowable Composite | Conventional Composite
Number analyzed (Participants) | 49 | 49
Number analyzed (teeth) | 49 | 49
units on a scale
  sensitiity to cold baseline | 1.6 (1.6) | 1.6 (2.0)
  sensitivity to biting baseline | 0.5 (0.6) | 0.7 (0.7)
  sensitiity to cold 6 Mo | 1.5 (1.4) | 1.8 (1.7)
  sensitiity to biting 6 Mo | 0.6 (0.7) | 0.8 (0.8)
  sensitiity to cold 12 Mo | 2.1 (2.2) | 1.7 (1.7)
  sensitiity to biting 12 Mo | 0.3 (0.5) | 0.3 (0.5)
  sensitiity to cold 24 Mo | 1.5 (1.9) | 1.0 (1.3)
  sensitiity to biting 24 Mo | 0.2 (0.5) | 0.1 (0.3)
Statistical Analysis 1: Comparison: Flowable Composite vs Conventional Composite; null hypothesis no difference in sensitivity to cold; Test type: Superiority or Other; p = 0.522, ANOVA
Statistical Analysis 2: Comparison: Flowable Composite vs Conventional Composite; null hypothesis no difference in biting pressure; Test type: Superiority or Other; p = .449, Chi-squared

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No